CLINICAL TRIAL: NCT01374178
Title: Relative Bioavailability of LY2963016 to LANTUS® After Single Dose Subcutaneous Administration to Healthy Subjects
Brief Title: A Comparison of LY2963016 to a Basal Insulin After a Single Dose in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14094; I4L-MC-ABEI (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — LY2963016 insulin glargine; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2963016 (Experimental): A single 0.5-unit per kilogram (U/kg) dose of LY2963016 will be administered subcutaneously.
  Interventions: Drug: LY2963016
- Lantus (Active Comparator): A single 0.5-U/kg dose of Lantus will be administered subcutaneously.
  Interventions: Drug: Lantus

INTERVENTIONS:
Drug: LY2963016 — Administered subcutaneously
  Arms: LY2963016
Drug: Lantus — Administered subcutaneously
  Other Names: Insulin Glargine
  Arms: Lantus

SUMMARY:
The purposes of this study are to determine the pharmacokinetics and pharmacodynamics of LY2963016 compared to those of basal insulin. The study will also gather information on the safety and tolerability of LY2963016 in healthy subjects. The study is approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females
* Have a body mass index (BMI) between 18.5 and 29.9 kilogram per square meter (kg/m^2)
* Are nonsmokers
* Have normal blood pressure and pulse rate
* Have an electrocardiogram (ECG) considered as within normal limits
* Have clinical laboratory test results within normal reference range

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device
* Have known allergies to insulin or its excipients
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Show evidence of significant active neuropsychiatric disease
* Have a history of first-degree relatives known to have diabetes mellitus
* Have a fasting venous blood glucose >6.0 millimoles per liter (mmol/L)
* Intend to use over-the-counter or prescription medication
* Have donated or had a blood loss of 450 milliliters (mL) or more in the past 3 months
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2963016 First, Then Lantus: A single 0.5-unit per kilogram (U/kg) dose of LY2963016 was administered subcutaneously during Period 1 (1 period=24 hours), followed by a washout period of at least 7 days before a single 0.5-U/kg Lantus dose was administered subcutaneously during Period 2 (1 period=24 hours).
- Lantus First, Then LY2963016: A single 0.5-U/kg dose of Lantus was administered subcutaneously during Period 1 (1 period=24 hours), followed by a washout period of at least 7 days before a single 0.5-U/kg dose of LY2963016 was administered subcutaneously during Period 2 (1 period=24 hours).
Period: Period 1 (up to 24 Hours After Dosing)
Arm/Group | LY2963016 First, Then Lantus | Lantus First, Then LY2963016
Started | 11 | 5
Received at Least 1 Dose of LY2963016 | 11 | 5
Completed | 11 | 5
Not Completed | 0 | 0
Period: Washout Period of at Least 7 Days
Arm/Group | LY2963016 First, Then Lantus | Lantus First, Then LY2963016
Started | 11 | 5
Completed | 10 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2 (up to 24 Hours After Dosing)
Arm/Group | LY2963016 First, Then Lantus | Lantus First, Then LY2963016
Started | 10 | 5
Completed | 8 | 5
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: For the LY2963016 first, then Lantus group: A single 0.5-unit per kilogram (U/kg) dose of LY2963016 was administered subcutaneously during Period 1 (1 period=24 hours), followed by a washout period of at least 7 days before a single 0.5-U/kg Lantus dose was administered subcutaneously during Period 2 (1 period=24 hours).
  For the Lantus first, then LY2963016 group: A single 0.5-U/kg dose of Lantus was administered subcutaneously during Period 1 (1 period=24 hours), followed by a washout period of at least 7 days before a single 0.5-U/kg dose of LY2963016 was administered subcutaneously during Period 2 (1 period=24 hours).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC)
Description: AUC from time zero to 24 hours (AUC0-24) is reported for this outcome measure.
Time Frame: Periods 1 and 2: Baseline up to 24 hours
Population: All randomized participants who received at least 1 dose of study drug, completed at least 1 clamp procedure, and had evaluable pharmacokinetic data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour per liter (pmol*hr/L)
Groups:
- LY2963016: A single 0.5-unit per kilogram (U/kg) dose of LY2963016 was administered subcutaneously.
- Lantus: A single 0.5-U/kg dose of Lantus was administered subcutaneously.
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 16 | 13
picomole*hour per liter (pmol*hr/L) | 1900 (22) | 2180 (30)

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax)
Time Frame: Periods 1 and 2: Baseline up to 24 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole per liter (pmol/L)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 16 | 13
picomole per liter (pmol/L) | 110 (26) | 130 (35)

3. Secondary Outcome: Maximum Glucose Infusion Rate (Rmax)
Time Frame: Periods 1 and 2: Baseline up to 24 hours
Population: All randomized participants who received at least 1 dose of study drug, completed at least 1 clamp procedure, and had evaluable glucodynamic data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams per hour (g/h)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 16 | 13
grams per hour (g/h) | 10.2 (50) | 11.3 (32)

4. Secondary Outcome: Total Glucose Infused (Gtot)
Time Frame: Periods 1 and 2: Baseline up to 24 hours
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: gram (g)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 16 | 13
gram (g) | 141 (54) | 160 (36)

5. Secondary Outcome: Time of Maximum Glucose Infusion Rate (tRmax)
Time Frame: Periods 1 and 2: Baseline up to 24 hours
Population: All randomized participants who received at least 1 dose of study drug, completed at least 1 clamp procedure, and had evaluable glucodynamic data.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 16 | 13
hour (h) | 10.5 [5.40 to 15.1] | 10.2 [5.50 to 15.8]

6. Secondary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects were defined as serious and nonserious adverse events. A summary of serious and all other nonserious adverse events is located in the Reported Adverse Event module.
Time Frame: Baseline up to 30 days
Population: All randomized participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 16 | 13
participants
  Serious Adverse Events | 0 | 0
  Nonserious Adverse Events | 8 | 6

ADVERSE EVENTS:
Arm/Group | LY2963016 | Lantus
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 8/16 | 6/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 (N=16) | Lantus (N=13)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 1 (1)
Catheter site swelling (General disorders) | 3 (3) | 1 (1)
Chest discomfort (General disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes